CLINICAL TRIAL: NCT05906628
Title: A Phase 2, Double-Blind, Randomized, 16-Week, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream Followed by an Open-Label Extension Period in Adults With Chronic Hand Eczema
Brief Title: Topical Ruxolitinib Evaluation in Chronic Hand Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 18424-226; 2022-502827-23-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Hand Eczema
Keywords: eczema; chronic hand eczema (CHE); dermatitis; skin disease; JAK inhibitor
MeSH Terms: conditions — Eczema; Dermatitis; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Participants will receive ruxolitinib cream (1.5%) or vehicle cream for 16 weeks, after which they will be offered the opportunity to receive ruxilitinib cream (1.5%) in the open-label treatment extension period for another 16 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib cream 1.5% twice daily (BID) for 16 weeks followed by ruxolitinib cream 1.5% BID for an additional 16-week treatment extension period.
  Interventions: Drug: Ruxolitinib cream
- Vehicle (Placebo Comparator): Vehicle cream for 16 weeks followed by crossover to ruxolitinib cream 1.5% BID in a 16-week treatment extension period.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Ruxolitinib cream — Ruxolitinib cream is a topical formulation applied as a thin film to affected areas.
  Other Names: INCB18424 cream
  Arms: Ruxolitinib
Drug: Vehicle — Vehicle cream is a topical formulation applied as a thin film to affected areas.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in adult participants with diagnosis of chronic hand eczema (CHE) and moderate to severe disease activity (Investigator's Global Assessement (IGA) of CHE score 3 or 4).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CHE for at least 6 months prior to screening. Diagnosis of chromic hand eczema (CHE) as defined by hand eczema (HE) lasting > 3 months or ≥ 2 flares within the previous 12 months.
* Screening and baseline IGA-CHE 3 or 4.
* Baseline CHE-related Itch NRS ≥ 4.
* Have been treated with at least 1 prescription CHE therapy or if such therapy was not advisable or contraindicated.
* Willingness to avoid pregnancy or fathering children based on the criteria defined in the protocol.

Exclusion Criteria:

* Known triggers for CHE (allergic or irritant, such as those identified by previous patch tests) cannot be avoided during the course of this study.
* Any serious illness or medical, physical, or psychiatric condition(s).
* Laboratory values outside of the protocol-defined criteria.
* Use of protocol-defined treatments within the indicated washout period before baseline.
* Psoralen ultraviolet A (PUVA) or ultraviolet B (UVB) therapy on the hands within 4 weeks before baseline.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (36):
- United States (23):
  - Southwest Skin Specialists Phoenix Biltmore, Phoenix, Arizona
  - First Oc Dermatology, Fountain Valley, California
  - Marvel Clinical Research Llc, Huntington Beach, California
  - Dermatology Research Associates, Los Angeles, California
  - Skin Research of South Florida, Llc, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Midwest Allergy Sinus Asthma, Sc, Normal, Illinois
  - The Indiana Clinical Trials Center Ictc, Plainfield, Indiana
  - Delricht Research, Baton Rouge, Louisiana
  - Delricht Research, New Orleans, Louisiana
  - Henry Ford Medical Center, Detroit, Michigan
  - Jubilee Clinical Research Inc, Las Vegas, Nevada
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Juva Skin and Laser Center, New York, New York
  - Onsite Clinical Solutions, Llc Charlotte Central Office, Charlotte, North Carolina
  - Bexley Dermatology, Bexley, Ohio
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Canada (3):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Care Clinic, Red Deer, Alberta
  - Simcomed Health Ltd, Barrie, Ontario
- Germany (4):
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim
  - Derma-Study-Center Fn Gmbh, Friedrichshafen
  - Dermatologische Gemeinschaftspraxis Mahlow, Mahlow
  - Beldio Research Gmbh, Memmingen
- Poland (6):
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp. Z O.O., Elblag
  - Centrum Badan Klinicznych Pi-House Sp. Z O.O., Gdansk
  - Laser Clinic S.C., Szczecin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Klinika Ambroziak, Warsaw
  - Dermmedica Sp. Z O.O., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 30 study centers in Canada, Germany, Poland, and the United States.
Groups:
- Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) to chronic hand eczema (CHE) lesions on the hands and wrists (if applicable) for 16 weeks. Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied ruxolitinib 1.5% cream BID during the DBVC Period continued to apply ruxolitinib 1.5% cream BID as needed for an additional 16 weeks in the OLE Period.
- Vehicle Cream BID to Ruxolitinib 1.5% Cream BID: Participants applied matching vehicle cream BID to CHE lesions on the hands and wrists (if applicable) for 16 weeks. Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied vehicle cream BID during the DBVC Period applied ruxolitinib 1.5% cream BID as needed for 16 weeks in the OLE Period.
Period: 16-Week DBVC Period
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Started | 94 | 92
Completed | 84 | 77
Not Completed | 10 | 15
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 4 | 11
Period: 16-Week OLE Period
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Started | 84 | 77
Completed | 76 | 71
Not Completed | 8 | 6
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Total
Number analyzed (Participants) | 94 | 92 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.11) | 48.1 (15.29) | 48.0 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 38 | 37 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 87 | 85 | 172
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 83 | 85 | 168
  Black/African American | 5 | 3 | 8
  Asian | 5 | 2 | 7
  Not Reported | 0 | 1 | 1
  Indian | 1 | 0 | 1
  Middle Eastern | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment-Chronic Hand Eczema Treatment Success (IGA-CHE-TS) at Week 16
Description: The Investigator's Global Assessment-Chronic Hand Eczema (IGA-CHE) is an instrument used to rate the severity of the participant's global CHE and is based on a 5-point scale ranging from 0 (clear) to 4 (severe) (1, almost clear; 2, mild eczema; 3, moderate eczema). IGA-CHE TS is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from Baseline.
Time Frame: Baseline; Week 16
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to the study. Treatment groups were defined according to the treatment assignment at the time of randomization regardless of the actual study treatment the participant might have applied during their participation in the study. Missing post-Baseline values were imputed as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
percentage of participants | 53.2 [42.6 to 63.6] | 10.9 [5.3 to 19.1]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test was stratified by stratification factors IGA-CHE score (3 or 4) and region (North America or outside of North America); Odds Ratio (OR) = 9.82, 95% CI 2-sided [4.48 to 21.49]
Statistical Analysis 2: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response rate difference = 42.5, 95% CI 2-sided [30.70 to 54.36], Standard Error of Mean 6.03

2. Secondary Outcome: Percentage of Participants Achieving ITCH4 Response at Weeks 4 and 16
Description: ITCH4 response was defined as a ≥4-point improvement in CHE-related Itch Numerical Rating Scale (NRS) score from Baseline. The CHE-related Itch NRS is a once-per-24 hours ("daily") participant-reported measure of the worst itch severity of their CHE assessed using an 11-point scale (0=no itch to 10=worst imaginable itch).
Time Frame: Baseline; Weeks 4 and 16
Population: ITT Population. Participants with a Baseline Itch NRS Score ≥4 were analyzed. Missing post-Baseline values were imputed as nonresponders at Weeks 4 and 16.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92 | 91
percentage of participants
  Week 4 | 46.7 [36.3 to 57.4] | 17.6 [10.4 to 27.0]
  Week 16 | 52.2 [41.5 to 62.7] | 23.1 [14.9 to 33.1]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.23, 95% CI 2-sided [2.14 to 8.38]
Statistical Analysis 2: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; Response rate difference = 29.5, 95% CI 2-sided [16.69 to 42.24], Standard Error of Mean 6.52
Statistical Analysis 3: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.90, 95% CI 2-sided [2.02 to 7.51]
Statistical Analysis 4: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 16; Test type: Superiority; Response rate difference = 29.5, 95% CI 2-sided [16.34 to 42.57], Standard Error of Mean 6.69

3. Secondary Outcome: Percentage of Participants Achieving ITCH4 Response at Day 3 and Week 1 (Day 7)
Description: as for outcome 2
Time Frame: Baseline; Day 3; Week 1 (Day 7)
Population: ITT Population. Participants with a Baseline Itch NRS Score ≥4 were analyzed. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 88 | 90
percentage of participants
  Day 3: number analyzed (Participants) | 85 | 83
  Day 3 | 12.9 [6.6 to 22.0] | 6.0 [2.0 to 13.5]
  Week 1 (Day 7): number analyzed (Participants) | 82 | 84
  Week 1 (Day 7) | 28.0 [18.7 to 39.1] | 9.5 [4.2 to 17.9]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Day 3; Test type: Superiority; p = 0.1789, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.718 to 5.923]
Statistical Analysis 2: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 1 (Day 7); Test type: Superiority; p = 0.0024, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.79, 95% CI 2-sided [1.603 to 8.951]

4. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment-Chronic Hand Eczema Treatment Success (IGA-CHE-TS) at Each Post-Baseline Visit
Description: The IGA-CHE is an instrument used to rate the severity of the participant's global CHE and is based on a 5-point scale ranging from 0 (clear) to 4 (severe) (1, almost clear; 2, mild eczema; 3, moderate eczema). IGA-CHE TS is defined as an IGA-CHE score of 0 (clear) or 1 (almost clear) with a ≥2-step improvement from Baseline.
Time Frame: Baseline; Weeks 2, 4, 8, 12, 16, 24, and 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
percentage of participants
  Week 2: number analyzed (Participants) | 89 | 86
  Week 2 | 22.5 [14.3 to 32.6] | 1.2 [0.0 to 6.3]
  Week 4: number analyzed (Participants) | 90 | 84
  Week 4 | 37.8 [27.8 to 48.6] | 4.8 [1.3 to 11.7]
  Week 8: number analyzed (Participants) | 88 | 80
  Week 8 | 44.3 [33.7 to 55.3] | 3.8 [0.8 to 10.6]
  Week 12: number analyzed (Participants) | 87 | 78
  Week 12 | 52.9 [41.9 to 63.7] | 14.1 [7.3 to 23.8]
  Week 16: number analyzed (Participants) | 86 | 78
  Week 16 | 58.1 [47.0 to 68.7] | 12.8 [6.3 to 22.3]
  Week 24: number analyzed (Participants) | 82 | 74
  Week 24 | 51.2 [39.9 to 62.4] | 51.4 [39.4 to 63.1]
  Week 32: number analyzed (Participants) | 78 | 73
  Week 32 | 52.6 [40.9 to 64.0] | 54.8 [42.7 to 66.5]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 16; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 9.91, 95% CI 2-sided [4.44 to 22.13]
Statistical Analysis 2: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Week 16; Test type: Superiority; Response rate difference = 45.6, 95% CI 2-sided [32.83 to 58.27], Standard Error of Mean 6.49

5. Secondary Outcome: Change From Baseline in CHE-related Itch NRS Score at Each Post-Baseline Visit
Description: The CHE-related Itch NRS is a once-per-24 hours ("daily") participant-reported measure of the worst itch severity of their CHE assessed using an 11-point scale (0=no itch to 10=worst imaginable itch). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 1-32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Baseline: number analyzed (Participants) | 93 | 91
  Baseline | 6.68 (1.619) | 6.63 (1.592)
  Change from Baseline at Week 2: number analyzed (Participants) | 85 | 84
  Change from Baseline at Week 2 | -3.03 (2.346) | -1.34 (1.725)
  Change from Baseline at Week 4: number analyzed (Participants) | 87 | 82
  Change from Baseline at Week 4 | -3.88 (2.275) | -2.02 (2.062)
  Change from Baseline at Week 8: number analyzed (Participants) | 83 | 77
  Change from Baseline at Week 8 | -4.23 (2.437) | -2.20 (2.353)
  Change from Baseline at Week 12: number analyzed (Participants) | 77 | 73
  Change from Baseline at Week 12 | -4.41 (2.315) | -2.51 (2.350)
  Change from Baseline at Week 16: number analyzed (Participants) | 74 | 72
  Change from Baseline at Week 16 | -4.24 (2.279) | -2.47 (2.226)
  Change from Baseline at Week 24: number analyzed (Participants) | 68 | 62
  Change from Baseline at Week 24 | -4.23 (2.400) | -4.85 (2.323)
  Change from Baseline at Week 32: number analyzed (Participants) | 68 | 62
  Change from Baseline at Week 32 | -4.41 (2.163) | -5.01 (2.095)

6. Secondary Outcome: Time to ≥4-point Improvement From Baseline in CHE-related Itch NRS Score
Description: as for outcome 2
Time Frame: Baseline; up to Week 32
Population: ITT Population. Participants with a Baseline Itch NRS Score ≥4 were analyzed. The 95% confidence interval was calculated based on the Brookmeyer and Crowley method.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 88 | 90
days | 15.0 [12.0 to 18.0] | 29.0 [17.0 to 73.0]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0025, Log Rank; stratified by randomization stratification factors; Cox regression model = 1.719, 95% CI 2-sided [1.211 to 2.440] — Cox regression model stratified by stratification factors (Baseline IGA-CHE 3/4, Region : North America or outside of North America) was conducted to compare the difference in hazard rate between treatment and vehicle

7. Secondary Outcome: Change From Baseline in CHE-related Pain NRS Score at Each Post-Baseline Visit
Description: The CHE-related Pain NRS is a once-per-24 hours ("daily") participant-reported measure of the worst pain severity of their CHE assessed using an 11-point scale (0=no pain to 10=worst imaginable pain). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Weeks 1-32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Baseline: number analyzed (Participants) | 93 | 91
  Baseline | 6.14 (2.164) | 6.06 (1.754)
  Change from Baseline at Week 2: number analyzed (Participants) | 85 | 84
  Change from Baseline at Week 2 | -2.86 (2.433) | -1.27 (1.671)
  Change from Baseline at Week 4: number analyzed (Participants) | 87 | 82
  Change from Baseline at Week 4 | -3.82 (2.435) | -1.83 (1.929)
  Change from Baseline at Week 8: number analyzed (Participants) | 83 | 77
  Change from Baseline at Week 8 | -4.15 (2.625) | -1.95 (2.118)
  Change from Baseline at Week 12: number analyzed (Participants) | 77 | 73
  Change from Baseline at Week 12 | -4.25 (2.415) | -2.21 (2.206)
  Change from Baseline at Week 16: number analyzed (Participants) | 74 | 72
  Change from Baseline at Week 16 | -4.23 (2.627) | -2.32 (2.036)
  Change from Baseline at Week 24: number analyzed (Participants) | 68 | 62
  Change from Baseline at Week 24 | -4.25 (2.584) | -4.47 (2.261)
  Change from Baseline at Week 32: number analyzed (Participants) | 69 | 62
  Change from Baseline at Week 32 | -4.37 (2.524) | -4.61 (2.112)

8. Secondary Outcome: Percentage of Participants Achieving ≥2-point Improvement in CHE-related Skin Pain NRS Score From Baseline to Week 16
Description: The CHE-related Pain NRS is a once-per-24 hours ("daily") participant-reported measure of the worst pain severity of their CHE assessed using an 11-point scale (0=no pain to 10=worst imaginable pain).
Time Frame: Baseline; up to Week 16
Population: ITT Population. Participants with a Baseline Pain NRS Score ≥2 were analyzed. Only participants with available data were analyzed. The 95% confidence interval was calculated using the method by Brookmeyer and Crowley.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 91 | 89
percentage of participants
  Week 2: number analyzed (Participants) | 83 | 82
  Week 2 | 59.0 [47.693 to 69.715] | 34.1 [24.027 to 45.449]
  Week 4: number analyzed (Participants) | 86 | 80
  Week 4 | 76.7 [66.394 to 85.179] | 47.5 [36.213 to 58.977]
  Week 8: number analyzed (Participants) | 82 | 75
  Week 8 | 74.4 [63.555 to 83.396] | 52.0 [40.151 to 63.686]
  Week 12: number analyzed (Participants) | 75 | 71
  Week 12 | 84.0 [73.719 to 91.450] | 53.5 [41.287 to 65.452]
  Week 16: number analyzed (Participants) | 72 | 70
  Week 16 | 81.9 [71.106 to 90.021] | 58.6 [46.166 to 70.228]
  Week 24: number analyzed (Participants) | 66 | 61
  Week 24 | 83.3 [72.133 to 91.375] | 90.2 [79.810 to 96.304]
  Week 32: number analyzed (Participants) | 68 | 60
  Week 32 | 86.8 [76.356 to 93.765] | 88.3 [77.428 to 95.179]

9. Secondary Outcome: Time to ≥2-point Improvement From Baseline in CHE-related Skin Pain NRS Score
Description: as for outcome 8
Time Frame: Baseline; up to Week 32
Population: ITT Population. Participants with a Baseline Pain NRS Score ≥2 were analyzed. The 95% confidence interval was calculated using the method by Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92 | 90
days | 5.0 [4.0 to 7.0] | 8.0 [5.0 to 12.0]
Statistical Analysis 1: Comparison: Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID vs Vehicle Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.1319, Log Rank; stratified by randomization stratification factors; Cox regression model = 1.279, 95% CI 2-sided [0.931 to 1.759] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Percentage Change in Hand Eczema Severity Index (HECSI) Score From Baseline to Week 16
Description: The HECSI divides the hand into 5 areas for assessment (fingertips, fingers [except the tips], palms, back of hands, and wrists). Each of the 5 areas of the hand are assessed separately for erythema, induration/papulation, vesicles, fissuring, scaling, and edema using the following scale: 0, no skin changes; 1, mild disease; 2, moderate disease; and 3, severe disease. To determine the HECSI score, the affected area for each location (total of both hands) is given a score from 0 to 4 (0, 0%; 1, 1%-25%; 2, 26%-50%; 3, 51%-75%; and 4, 76%-100%) based on the extent of clinical symptoms. Finally, the score given for the extent at each location is multiplied by the total sum of the intensity of each clinical feature to calculate the total HECSI score, varying from 0 to a maximum severity score of 360 points. Percentage change was calculated as the ([post-Baseline value minus the Baseline value]/[Baseline value]) * 100.
Time Frame: Baseline; up to Week 16
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 92 | 90
percentage change
  Week 2: number analyzed (Participants) | 89 | 86
  Week 2 | -54.93 (34.148) | -16.68 (50.066)
  Week 4: number analyzed (Participants) | 90 | 84
  Week 4 | -69.58 (37.852) | -26.00 (58.790)
  Week 8: number analyzed (Participants) | 88 | 80
  Week 8 | -77.25 (29.583) | -33.81 (62.468)
  Week 12: number analyzed (Participants) | 87 | 78
  Week 12 | -78.65 (37.390) | -41.00 (50.605)
  Week 16: number analyzed (Participants) | 86 | 78
  Week 16 | -84.88 (22.971) | -37.61 (54.760)

11. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Each Post-Baseline Visit
Description: The PGIC is a participants' self-reporting measure that reflects their belief about the efficacy of treatment. The PGIC is a 7-point scale depicting a participant's rating of overall improvement of CHE. Participants were asked to select 1 response from the response options that best described the overall change in their CHE since they started study treatment: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse, and 7, very much worse.
Time Frame: Baseline; up to Week 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Week 2: number analyzed (Participants) | 88 | 84
  Week 2 | 1.85 (0.824) | 3.21 (1.309)
  Week 4: number analyzed (Participants) | 86 | 82
  Week 4 | 1.74 (0.897) | 3.09 (1.288)
  Week 8: number analyzed (Participants) | 85 | 79
  Week 8 | 1.64 (0.784) | 3.04 (1.344)
  Week 12: number analyzed (Participants) | 80 | 76
  Week 12 | 1.60 (0.851) | 3.04 (1.399)
  Week 16: number analyzed (Participants) | 80 | 77
  Week 16 | 1.61 (0.893) | 3.00 (1.308)
  Week 24: number analyzed (Participants) | 76 | 70
  Week 24 | 1.61 (0.750) | 1.73 (0.931)
  Week 32: number analyzed (Participants) | 72 | 67
  Week 32 | 1.57 (0.932) | 1.67 (0.877)

12. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Weeks 2, 4, 8, 12, 16, 24, and 32
Description: The DLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. The questionnaire was analyzed under 6 subscales as follows: symptoms and feelings (Questions 1 and 2); daily activities (Questions 3 and 4); leisure (Questions 5 and 6); work and school (Question 7); personal relations (Questions 8 and 9); and treatment (Question 10). Scoring of each question is as follows: very much = 3; a lot = 2; a little = 1; not at all = 0; not relevant = 0 (Question 7: "Prevented work or studying" = Yes = 3). The DLQI was calculated by summing the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life was impaired.
Time Frame: Baseline; up to Week 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Baseline: number analyzed (Participants) | 90 | 91
  Baseline | 13.17 (6.277) | 11.84 (5.896)
  Change from Baseline at Week 2: number analyzed (Participants) | 83 | 84
  Change from Baseline at Week 2 | -7.95 (5.046) | -3.62 (4.065)
  Change from Baseline at Week 4: number analyzed (Participants) | 82 | 82
  Change from Baseline at Week 4 | -8.68 (5.517) | -4.78 (5.116)
  Change from Baseline at Week 8: number analyzed (Participants) | 81 | 78
  Change from Baseline at Week 8 | -9.11 (5.837) | -5.32 (4.977)
  Change from Baseline at Week 12: number analyzed (Participants) | 77 | 75
  Change from Baseline at Week 12 | -9.38 (5.905) | -5.88 (5.964)
  Change from Baseline at Week 16: number analyzed (Participants) | 76 | 77
  Change from Baseline at Week 16 | -9.62 (6.055) | -5.36 (5.441)
  Change from Baseline at Week 24: number analyzed (Participants) | 73 | 70
  Change from Baseline at Week 24 | -8.97 (6.457) | -8.71 (5.517)
  Change from Baseline at Week 32: number analyzed (Participants) | 69 | 67
  Change from Baseline at Week 32 | -9.71 (5.675) | -9.34 (5.550)

13. Secondary Outcome: Number of Participants With the Indicated EQ-5D-5L Dimension Scores at Weeks 2, 4, 8, 12, 16, 24, and 32
Description: The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome. The EQ-5D-5L questionnaire consists of the following 2 sections: the EQ-5D descriptive system and the EQ Visual Analog Scale (VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: Level 1 = no problems; Level 2 = slight problems; Level 3 = moderate problems; Level 4 = severe problems; and Level 5 = extreme problems. The EQ VAS records the participant's self-rated health on a vertical VAS (0-100), where the endpoints are labeled "the best health you can imagine" (100 score) and "the worst health you can imagine" (0 score).
Time Frame: Baseline; up to Week 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
Participants
  Mobility; Baseline, Level 1: number analyzed (Participants) | 89 | 90
  Mobility; Baseline, Level 1 | 70 | 73
  Mobility; Baseline, Level 2: number analyzed (Participants) | 89 | 90
  Mobility; Baseline, Level 2 | 14 | 8
  Mobility; Baseline, Level 3: number analyzed (Participants) | 89 | 90
  Mobility; Baseline, Level 3 | 5 | 6
  Mobility; Baseline, Level 4: number analyzed (Participants) | 89 | 90
  Mobility; Baseline, Level 4 | 0 | 1
  Mobility; Baseline, Level 5: number analyzed (Participants) | 89 | 90
  Mobility; Baseline, Level 5 | 0 | 2
  Mobility; Week 2, Level 1: number analyzed (Participants) | 86 | 84
  Mobility; Week 2, Level 1 | 74 | 70
  Mobility; Week 2, Level 2: number analyzed (Participants) | 86 | 84
  Mobility; Week 2, Level 2 | 4 | 9
  Mobility; Week 2, Level 3: number analyzed (Participants) | 86 | 84
  Mobility; Week 2, Level 3 | 4 | 4
  Mobility; Week 2, Level 4: number analyzed (Participants) | 86 | 84
  Mobility; Week 2, Level 4 | 2 | 1
  Mobility; Week 2, Level 5: number analyzed (Participants) | 86 | 84
  Mobility; Week 2, Level 5 | 2 | 0
  Mobility; Week 4, Level 1: number analyzed (Participants) | 86 | 82
  Mobility; Week 4, Level 1 | 69 | 68
  Mobility; Week 4, Level 2: number analyzed (Participants) | 86 | 82
  Mobility; Week 4, Level 2 | 13 | 9
  Mobility; Week 4, Level 3: number analyzed (Participants) | 86 | 82
  Mobility; Week 4, Level 3 | 4 | 3
  Mobility; Week 4, Level 4: number analyzed (Participants) | 86 | 82
  Mobility; Week 4, Level 4 | 0 | 2
  Mobility; Week 4, Level 5: number analyzed (Participants) | 86 | 82
  Mobility; Week 4, Level 5 | 0 | 0
  Mobility; Week 8, Level 1: number analyzed (Participants) | 85 | 78
  Mobility; Week 8, Level 1 | 71 | 70
  Mobility; Week 8, Level 2: number analyzed (Participants) | 85 | 78
  Mobility; Week 8, Level 2 | 14 | 5
  Mobility; Week 8, Level 3: number analyzed (Participants) | 85 | 78
  Mobility; Week 8, Level 3 | 0 | 2
  Mobility; Week 8, Level 4: number analyzed (Participants) | 85 | 78
  Mobility; Week 8, Level 4 | 0 | 1
  Mobility; Week 8, Level 5: number analyzed (Participants) | 85 | 78
  Mobility; Week 8, Level 5 | 0 | 0
  Mobility; Week 12, Level 1: number analyzed (Participants) | 80 | 75
  Mobility; Week 12, Level 1 | 67 | 63
  Mobility; Week 12, Level 2: number analyzed (Participants) | 80 | 75
  Mobility; Week 12, Level 2 | 7 | 9
  Mobility; Week 12, Level 3: number analyzed (Participants) | 80 | 75
  Mobility; Week 12, Level 3 | 5 | 2
  Mobility; Week 12, Level 4: number analyzed (Participants) | 80 | 75
  Mobility; Week 12, Level 4 | 1 | 1
  Mobility; Week 12, Level 5: number analyzed (Participants) | 80 | 75
  Mobility; Week 12, Level 5 | 0 | 0
  Mobility; Week 16, Level 1: number analyzed (Participants) | 80 | 77
  Mobility; Week 16, Level 1 | 69 | 64
  Mobility; Week 16, Level 2: number analyzed (Participants) | 80 | 77
  Mobility; Week 16, Level 2 | 7 | 9
  Mobility; Week 16, Level 3: number analyzed (Participants) | 80 | 77
  Mobility; Week 16, Level 3 | 4 | 2
  Mobility; Week 16, Level 4: number analyzed (Participants) | 80 | 77
  Mobility; Week 16, Level 4 | 0 | 2
  Mobility; Week 16, Level 5: number analyzed (Participants) | 80 | 77
  Mobility; Week 16, Level 5 | 0 | 0
  Mobility; Week 24, Level 1: number analyzed (Participants) | 76 | 70
  Mobility; Week 24, Level 1 | 65 | 60
  Mobility; Week 24, Level 2: number analyzed (Participants) | 76 | 70
  Mobility; Week 24, Level 2 | 6 | 8
  Mobility; Week 24, Level 3: number analyzed (Participants) | 76 | 70
  Mobility; Week 24, Level 3 | 4 | 2
  Mobility; Week 24, Level 4: number analyzed (Participants) | 76 | 70
  Mobility; Week 24, Level 4 | 1 | 0
  Mobility; Week 24, Level 5: number analyzed (Participants) | 76 | 70
  Mobility; Week 24, Level 5 | 0 | 0
  Mobility; Week 32, Level 1: number analyzed (Participants) | 69 | 67
  Mobility; Week 32, Level 1 | 61 | 55
  Mobility; Week 32, Level 2: number analyzed (Participants) | 69 | 67
  Mobility; Week 32, Level 2 | 5 | 7
  Mobility; Week 32, Level 3: number analyzed (Participants) | 69 | 67
  Mobility; Week 32, Level 3 | 3 | 4
  Mobility; Week 32, Level 4: number analyzed (Participants) | 69 | 67
  Mobility; Week 32, Level 4 | 0 | 1
  Mobility; Week 32, Level 5: number analyzed (Participants) | 69 | 67
  Mobility; Week 32, Level 5 | 0 | 0
  Self-care; Baseline, Level 1: number analyzed (Participants) | 89 | 90
  Self-care; Baseline, Level 1 | 55 | 61
  Self-care; Baseline, Level 2: number analyzed (Participants) | 89 | 90
  Self-care; Baseline, Level 2 | 24 | 21
  Self-care; Baseline, Level 3: number analyzed (Participants) | 89 | 90
  Self-care; Baseline, Level 3 | 5 | 6
  Self-care; Baseline, Level 4: number analyzed (Participants) | 89 | 90
  Self-care; Baseline, Level 4 | 5 | 2
  Self-care; Baseline, Level 5: number analyzed (Participants) | 89 | 90
  Self-care; Baseline, Level 5 | 0 | 0
  Self-care; Week 2, Level 1: number analyzed (Participants) | 86 | 84
  Self-care; Week 2, Level 1 | 73 | 64
  Self-care; Week 2, Level 2: number analyzed (Participants) | 86 | 84
  Self-care; Week 2, Level 2 | 10 | 13
  Self-care; Week 2, Level 3: number analyzed (Participants) | 86 | 84
  Self-care; Week 2, Level 3 | 3 | 5
  Self-care; Week 2, Level 4: number analyzed (Participants) | 86 | 84
  Self-care; Week 2, Level 4 | 0 | 1
  Self-care; Week 2, Level 5: number analyzed (Participants) | 86 | 84
  Self-care; Week 2, Level 5 | 0 | 1
  Self-care; Week 4, Level 1: number analyzed (Participants) | 86 | 82
  Self-care; Week 4, Level 1 | 69 | 57
  Self-care; Week 4, Level 2: number analyzed (Participants) | 86 | 82
  Self-care; Week 4, Level 2 | 14 | 19
  Self-care; Week 4, Level 3: number analyzed (Participants) | 86 | 82
  Self-care; Week 4, Level 3 | 3 | 5
  Self-care; Week 4, Level 4: number analyzed (Participants) | 86 | 82
  Self-care; Week 4, Level 4 | 0 | 1
  Self-care; Week 4, Level 5: number analyzed (Participants) | 86 | 82
  Self-care; Week 4, Level 5 | 0 | 0
  Self-care; Week 8, Level 1: number analyzed (Participants) | 85 | 78
  Self-care; Week 8, Level 1 | 76 | 57
  Self-care; Week 8, Level 2: number analyzed (Participants) | 85 | 78
  Self-care; Week 8, Level 2 | 6 | 15
  Self-care; Week 8, Level 3: number analyzed (Participants) | 85 | 78
  Self-care; Week 8, Level 3 | 3 | 6
  Self-care; Week 8, Level 4: number analyzed (Participants) | 85 | 78
  Self-care; Week 8, Level 4 | 0 | 0
  Self-care; Week 8, Level 5: number analyzed (Participants) | 85 | 78
  Self-care; Week 8, Level 5 | 0 | 0
  Self-care; Week 12, Level 1: number analyzed (Participants) | 80 | 75
  Self-care; Week 12, Level 1 | 72 | 61
  Self-care; Week 12, Level 2: number analyzed (Participants) | 80 | 75
  Self-care; Week 12, Level 2 | 8 | 10
  Self-care; Week 12, Level 3: number analyzed (Participants) | 80 | 75
  Self-care; Week 12, Level 3 | 0 | 4
  Self-care; Week 12, Level 4: number analyzed (Participants) | 80 | 75
  Self-care; Week 12, Level 4 | 0 | 0
  Self-care; Week 12, Level 5: number analyzed (Participants) | 80 | 75
  Self-care; Week 12, Level 5 | 0 | 0
  Self-care; Week 16, Level 1: number analyzed (Participants) | 80 | 77
  Self-care; Week 16, Level 1 | 72 | 59
  Self-care; Week 16, Level 2: number analyzed (Participants) | 80 | 77
  Self-care; Week 16, Level 2 | 8 | 16
  Self-care; Week 16, Level 3: number analyzed (Participants) | 80 | 77
  Self-care; Week 16, Level 3 | 0 | 2
  Self-care; Week 16, Level 4: number analyzed (Participants) | 80 | 77
  Self-care; Week 16, Level 4 | 0 | 0
  Self-care; Week 16, Level 5: number analyzed (Participants) | 80 | 77
  Self-care; Week 16, Level 5 | 0 | 0
  Self-care; Week 24, Level 1: number analyzed (Participants) | 76 | 70
  Self-care; Week 24, Level 1 | 70 | 64
  Self-care; Week 24, Level 2: number analyzed (Participants) | 76 | 70
  Self-care; Week 24, Level 2 | 4 | 4
  Self-care; Week 24, Level 3: number analyzed (Participants) | 76 | 70
  Self-care; Week 24, Level 3 | 1 | 2
  Self-care; Week 24, Level 4: number analyzed (Participants) | 76 | 70
  Self-care; Week 24, Level 4 | 1 | 0
  Self-care; Week 24, Level 5: number analyzed (Participants) | 76 | 70
  Self-care; Week 24, Level 5 | 0 | 0
  Self-care; Week 32, Level 1: number analyzed (Participants) | 69 | 67
  Self-care; Week 32, Level 1 | 64 | 62
  Self-care; Week 32, Level 2: number analyzed (Participants) | 69 | 67
  Self-care; Week 32, Level 2 | 3 | 5
  Self-care; Week 32, Level 3: number analyzed (Participants) | 69 | 67
  Self-care; Week 32, Level 3 | 2 | 0
  Self-care; Week 32, Level 4: number analyzed (Participants) | 69 | 67
  Self-care; Week 32, Level 4 | 0 | 0
  Self-care; Week 32, Level 5: number analyzed (Participants) | 69 | 67
  Self-care; Week 32, Level 5 | 0 | 0
  Usual activities; Baseline, Level 1: number analyzed (Participants) | 89 | 90
  Usual activities; Baseline, Level 1 | 25 | 38
  Usual activities; Baseline, Level 2: number analyzed (Participants) | 89 | 90
  Usual activities; Baseline, Level 2 | 39 | 28
  Usual activities; Baseline, Level 3: number analyzed (Participants) | 89 | 90
  Usual activities; Baseline, Level 3 | 16 | 18
  Usual activities; Baseline, Level 4: number analyzed (Participants) | 89 | 90
  Usual activities; Baseline, Level 4 | 8 | 5
  Usual activities; Baseline, Level 5: number analyzed (Participants) | 89 | 90
  Usual activities; Baseline, Level 5 | 1 | 1
  Usual activities; Week 2, Level 1: number analyzed (Participants) | 86 | 84
  Usual activities; Week 2, Level 1 | 51 | 37
  Usual activities; Week 2, Level 2: number analyzed (Participants) | 86 | 84
  Usual activities; Week 2, Level 2 | 27 | 32
  Usual activities; Week 2, Level 3: number analyzed (Participants) | 86 | 84
  Usual activities; Week 2, Level 3 | 6 | 11
  Usual activities; Week 2, Level 4: number analyzed (Participants) | 86 | 84
  Usual activities; Week 2, Level 4 | 2 | 4
  Usual activities; Week 2, Level 5: number analyzed (Participants) | 86 | 84
  Usual activities; Week 2, Level 5 | 0 | 0
  Usual activities; Week 4, Level 1: number analyzed (Participants) | 86 | 82
  Usual activities; Week 4, Level 1 | 53 | 42
  Usual activities; Week 4, Level 2: number analyzed (Participants) | 86 | 82
  Usual activities; Week 4, Level 2 | 27 | 24
  Usual activities; Week 4, Level 3: number analyzed (Participants) | 86 | 82
  Usual activities; Week 4, Level 3 | 6 | 14
  Usual activities; Week 4, Level 4: number analyzed (Participants) | 86 | 82
  Usual activities; Week 4, Level 4 | 0 | 2
  Usual activities; Week 4, Level 5: number analyzed (Participants) | 86 | 82
  Usual activities; Week 4, Level 5 | 0 | 0
  Usual activities; Week 8, Level 1: number analyzed (Participants) | 85 | 78
  Usual activities; Week 8, Level 1 | 65 | 47
  Usual activities; Week 8, Level 2: number analyzed (Participants) | 85 | 78
  Usual activities; Week 8, Level 2 | 18 | 22
  Usual activities; Week 8, Level 3: number analyzed (Participants) | 85 | 78
  Usual activities; Week 8, Level 3 | 2 | 6
  Usual activities; Week 8, Level 4: number analyzed (Participants) | 85 | 78
  Usual activities; Week 8, Level 4 | 0 | 3
  Usual activities; Week 8, Level 5: number analyzed (Participants) | 85 | 78
  Usual activities; Week 8, Level 5 | 0 | 0
  Usual activities; Week 12, Level 1: number analyzed (Participants) | 80 | 75
  Usual activities; Week 12, Level 1 | 60 | 45
  Usual activities; Week 12, Level 2: number analyzed (Participants) | 80 | 75
  Usual activities; Week 12, Level 2 | 17 | 26
  Usual activities; Week 12, Level 3: number analyzed (Participants) | 80 | 75
  Usual activities; Week 12, Level 3 | 3 | 1
  Usual activities; Week 12, Level 4: number analyzed (Participants) | 80 | 75
  Usual activities; Week 12, Level 4 | 0 | 3
  Usual activities; Week 12, Level 5: number analyzed (Participants) | 80 | 75
  Usual activities; Week 12, Level 5 | 0 | 0
  Usual activities; Week 16, Level 1: number analyzed (Participants) | 80 | 77
  Usual activities; Week 16, Level 1 | 61 | 42
  Usual activities; Week 16, Level 2: number analyzed (Participants) | 80 | 77
  Usual activities; Week 16, Level 2 | 16 | 25
  Usual activities; Week 16, Level 3: number analyzed (Participants) | 80 | 77
  Usual activities; Week 16, Level 3 | 3 | 8
  Usual activities; Week 16, Level 4: number analyzed (Participants) | 80 | 77
  Usual activities; Week 16, Level 4 | 0 | 1
  Usual activities; Week 16, Level 5: number analyzed (Participants) | 80 | 77
  Usual activities; Week 16, Level 5 | 0 | 1
  Usual activities; Week 24, Level 1: number analyzed (Participants) | 76 | 70
  Usual activities; Week 24, Level 1 | 55 | 54
  Usual activities; Week 24, Level 2: number analyzed (Participants) | 76 | 70
  Usual activities; Week 24, Level 2 | 18 | 13
  Usual activities; Week 24, Level 3: number analyzed (Participants) | 76 | 70
  Usual activities; Week 24, Level 3 | 2 | 3
  Usual activities; Week 24, Level 4: number analyzed (Participants) | 76 | 70
  Usual activities; Week 24, Level 4 | 1 | 0
  Usual activities; Week 24, Level 5 | 0 | 0
  Usual activities; Week 32, Level 1: number analyzed (Participants) | 69 | 67
  Usual activities; Week 32, Level 1 | 57 | 61
  Usual activities; Week 32, Level 2: number analyzed (Participants) | 69 | 67
  Usual activities; Week 32, Level 2 | 8 | 4
  Usual activities; Week 32, Level 3: number analyzed (Participants) | 69 | 67
  Usual activities; Week 32, Level 3 | 4 | 2
  Usual activities; Week 32, Level 4: number analyzed (Participants) | 69 | 67
  Usual activities; Week 32, Level 4 | 0 | 0
  Usual activities; Week 32, Level 5: number analyzed (Participants) | 69 | 67
  Usual activities; Week 32, Level 5 | 0 | 0
  Pain/discomfort; Baseline, Level 1: number analyzed (Participants) | 89 | 90
  Pain/discomfort; Baseline, Level 1 | 3 | 5
  Pain/discomfort; Baseline, Level 2: number analyzed (Participants) | 89 | 90
  Pain/discomfort; Baseline, Level 2 | 28 | 28
  Pain/discomfort; Baseline, Level 3: number analyzed (Participants) | 89 | 90
  Pain/discomfort; Baseline, Level 3 | 37 | 36
  Pain/discomfort; Baseline, Level 4: number analyzed (Participants) | 89 | 90
  Pain/discomfort; Baseline, Level 4 | 20 | 19
  Pain/discomfort; Baseline, Level 5: number analyzed (Participants) | 89 | 90
  Pain/discomfort; Baseline, Level 5 | 1 | 2
  Pain/discomfort; Week 2, Level 1: number analyzed (Participants) | 86 | 84
  Pain/discomfort; Week 2, Level 1 | 33 | 17
  Pain/discomfort; Week 2, Level 2: number analyzed (Participants) | 86 | 84
  Pain/discomfort; Week 2, Level 2 | 37 | 35
  Pain/discomfort; Week 2, Level 3: number analyzed (Participants) | 86 | 84
  Pain/discomfort; Week 2, Level 3 | 14 | 20
  Pain/discomfort; Week 2, Level 4: number analyzed (Participants) | 86 | 84
  Pain/discomfort; Week 2, Level 4 | 2 | 11
  Pain/discomfort; Week 2, Level 5: number analyzed (Participants) | 86 | 84
  Pain/discomfort; Week 2, Level 5 | 0 | 1
  Pain/discomfort; Week 4, Level 1: number analyzed (Participants) | 86 | 82
  Pain/discomfort; Week 4, Level 1 | 37 | 15
  Pain/discomfort; Week 4, Level 2: number analyzed (Participants) | 86 | 82
  Pain/discomfort; Week 4, Level 2 | 38 | 38
  Pain/discomfort; Week 4, Level 3: number analyzed (Participants) | 86 | 82
  Pain/discomfort; Week 4, Level 3 | 9 | 25
  Pain/discomfort; Week 4, Level 4: number analyzed (Participants) | 86 | 82
  Pain/discomfort; Week 4, Level 4 | 2 | 2
  Pain/discomfort; Week 4, Level 5: number analyzed (Participants) | 86 | 82
  Pain/discomfort; Week 4, Level 5 | 0 | 2
  Pain/discomfort; Week 8, Level 1: number analyzed (Participants) | 85 | 78
  Pain/discomfort; Week 8, Level 1 | 46 | 22
  Pain/discomfort; Week 8, Level 2: number analyzed (Participants) | 85 | 78
  Pain/discomfort; Week 8, Level 2 | 29 | 36
  Pain/discomfort; Week 8, Level 3: number analyzed (Participants) | 85 | 78
  Pain/discomfort; Week 8, Level 3 | 10 | 13
  Pain/discomfort; Week 8, Level 4: number analyzed (Participants) | 85 | 78
  Pain/discomfort; Week 8, Level 4 | 0 | 7
  Pain/discomfort; Week 8, Level 5: number analyzed (Participants) | 85 | 78
  Pain/discomfort; Week 8, Level 5 | 0 | 0
  Pain/discomfort; Week 12, Level 1: number analyzed (Participants) | 80 | 75
  Pain/discomfort; Week 12, Level 1 | 40 | 20
  Pain/discomfort; Week 12, Level 2: number analyzed (Participants) | 80 | 75
  Pain/discomfort; Week 12, Level 2 | 30 | 37
  Pain/discomfort; Week 12, Level 3: number analyzed (Participants) | 80 | 75
  Pain/discomfort; Week 12, Level 3 | 9 | 16
  Pain/discomfort; Week 12, Level 4: number analyzed (Participants) | 80 | 75
  Pain/discomfort; Week 12, Level 4 | 1 | 1
  Pain/discomfort; Week 12, Level 5: number analyzed (Participants) | 80 | 75
  Pain/discomfort; Week 12, Level 5 | 0 | 1
  Pain/discomfort; Week 16, Level 1: number analyzed (Participants) | 80 | 77
  Pain/discomfort; Week 16, Level 1 | 42 | 20
  Pain/discomfort; Week 16, Level 2: number analyzed (Participants) | 80 | 77
  Pain/discomfort; Week 16, Level 2 | 28 | 38
  Pain/discomfort; Week 16, Level 3: number analyzed (Participants) | 80 | 77
  Pain/discomfort; Week 16, Level 3 | 6 | 14
  Pain/discomfort; Week 16, Level 4: number analyzed (Participants) | 80 | 77
  Pain/discomfort; Week 16, Level 4 | 4 | 4
  Pain/discomfort; Week 16, Level 5: number analyzed (Participants) | 80 | 77
  Pain/discomfort; Week 16, Level 5 | 0 | 1
  Pain/discomfort; Week 24, Level 1: number analyzed (Participants) | 76 | 70
  Pain/discomfort; Week 24, Level 1 | 42 | 40
  Pain/discomfort; Week 24, Level 2: number analyzed (Participants) | 76 | 70
  Pain/discomfort; Week 24, Level 2 | 26 | 22
  Pain/discomfort; Week 24, Level 3: number analyzed (Participants) | 76 | 70
  Pain/discomfort; Week 24, Level 3 | 7 | 7
  Pain/discomfort; Week 24, Level 4: number analyzed (Participants) | 76 | 70
  Pain/discomfort; Week 24, Level 4 | 0 | 1
  Pain/discomfort; Week 24, Level 5: number analyzed (Participants) | 76 | 70
  Pain/discomfort; Week 24, Level 5 | 1 | 0
  Pain/discomfort; Week 32, Level 1: number analyzed (Participants) | 69 | 67
  Pain/discomfort; Week 32, Level 1 | 35 | 39
  Pain/discomfort; Week 32, Level 2: number analyzed (Participants) | 69 | 67
  Pain/discomfort; Week 32, Level 2 | 27 | 22
  Pain/discomfort; Week 32, Level 3: number analyzed (Participants) | 69 | 67
  Pain/discomfort; Week 32, Level 3 | 7 | 5
  Pain/discomfort; Week 32, Level 4: number analyzed (Participants) | 69 | 67
  Pain/discomfort; Week 32, Level 4 | 0 | 1
  Pain/discomfort; Week 32, Level 5: number analyzed (Participants) | 69 | 67
  Pain/discomfort; Week 32, Level 5 | 0 | 0
  Anxiety/depression; Baseline, Level 1: number analyzed (Participants) | 89 | 90
  Anxiety/depression; Baseline, Level 1 | 39 | 41
  Anxiety/depression; Baseline, Level 2: number analyzed (Participants) | 89 | 90
  Anxiety/depression; Baseline, Level 2 | 28 | 28
  Anxiety/depression; Baseline, Level 3: number analyzed (Participants) | 89 | 90
  Anxiety/depression; Baseline, Level 3 | 16 | 11
  Anxiety/depression; Baseline, Level 4: number analyzed (Participants) | 89 | 90
  Anxiety/depression; Baseline, Level 4 | 5 | 9
  Anxiety/depression; Baseline, Level 5: number analyzed (Participants) | 89 | 90
  Anxiety/depression; Baseline, Level 5 | 1 | 1
  Anxiety/depression; Week 2, Level 1: number analyzed (Participants) | 86 | 84
  Anxiety/depression; Week 2, Level 1 | 56 | 43
  Anxiety/depression; Week 2, Level 2: number analyzed (Participants) | 86 | 84
  Anxiety/depression; Week 2, Level 2 | 22 | 29
  Anxiety/depression; Week 2, Level 3: number analyzed (Participants) | 86 | 84
  Anxiety/depression; Week 2, Level 3 | 6 | 8
  Anxiety/depression; Week 2, Level 4: number analyzed (Participants) | 86 | 84
  Anxiety/depression; Week 2, Level 4 | 2 | 3
  Anxiety/depression; Week 2, Level 5: number analyzed (Participants) | 86 | 84
  Anxiety/depression; Week 2, Level 5 | 0 | 1
  Anxiety/depression; Week 4, Level 1: number analyzed (Participants) | 86 | 82
  Anxiety/depression; Week 4, Level 1 | 53 | 46
  Anxiety/depression; Week 4, Level 2: number analyzed (Participants) | 86 | 82
  Anxiety/depression; Week 4, Level 2 | 24 | 24
  Anxiety/depression; Week 4, Level 3: number analyzed (Participants) | 86 | 82
  Anxiety/depression; Week 4, Level 3 | 7 | 6
  Anxiety/depression; Week 4, Level 4: number analyzed (Participants) | 86 | 82
  Anxiety/depression; Week 4, Level 4 | 2 | 5
  Anxiety/depression; Week 4, Level 5: number analyzed (Participants) | 86 | 82
  Anxiety/depression; Week 4, Level 5 | 0 | 1
  Anxiety/depression; Week 8, Level 1: number analyzed (Participants) | 85 | 78
  Anxiety/depression; Week 8, Level 1 | 57 | 46
  Anxiety/depression; Week 8, Level 2: number analyzed (Participants) | 85 | 78
  Anxiety/depression; Week 8, Level 2 | 23 | 24
  Anxiety/depression; Week 8, Level 3: number analyzed (Participants) | 85 | 78
  Anxiety/depression; Week 8, Level 3 | 3 | 5
  Anxiety/depression; Week 8, Level 4: number analyzed (Participants) | 85 | 78
  Anxiety/depression; Week 8, Level 4 | 1 | 3
  Anxiety/depression; Week 8, Level 5: number analyzed (Participants) | 85 | 78
  Anxiety/depression; Week 8, Level 5 | 1 | 0
  Anxiety/depression; Week 12, Level 1: number analyzed (Participants) | 80 | 75
  Anxiety/depression; Week 12, Level 1 | 58 | 46
  Anxiety/depression; Week 12, Level 2: number analyzed (Participants) | 80 | 75
  Anxiety/depression; Week 12, Level 2 | 15 | 19
  Anxiety/depression; Week 12, Level 3: number analyzed (Participants) | 80 | 75
  Anxiety/depression; Week 12, Level 3 | 5 | 7
  Anxiety/depression; Week 12, Level 4: number analyzed (Participants) | 80 | 75
  Anxiety/depression; Week 12, Level 4 | 1 | 2
  Anxiety/depression; Week 12, Level 5: number analyzed (Participants) | 80 | 75
  Anxiety/depression; Week 12, Level 5 | 1 | 1
  Anxiety/depression; Week 16, Level 1: number analyzed (Participants) | 80 | 77
  Anxiety/depression; Week 16, Level 1 | 54 | 46
  Anxiety/depression; Week 16, Level 2: number analyzed (Participants) | 80 | 77
  Anxiety/depression; Week 16, Level 2 | 19 | 23
  Anxiety/depression; Week 16, Level 3: number analyzed (Participants) | 80 | 77
  Anxiety/depression; Week 16, Level 3 | 4 | 5
  Anxiety/depression; Week 16, Level 4: number analyzed (Participants) | 80 | 77
  Anxiety/depression; Week 16, Level 4 | 3 | 2
  Anxiety/depression; Week 16, Level 5: number analyzed (Participants) | 80 | 77
  Anxiety/depression; Week 16, Level 5 | 0 | 1
  Anxiety/depression; Week 24, Level 1: number analyzed (Participants) | 76 | 70
  Anxiety/depression; Week 24, Level 1 | 54 | 50
  Anxiety/depression; Week 24, Level 2: number analyzed (Participants) | 76 | 70
  Anxiety/depression; Week 24, Level 2 | 17 | 15
  Anxiety/depression; Week 24, Level 3: number analyzed (Participants) | 76 | 70
  Anxiety/depression; Week 24, Level 3 | 3 | 3
  Anxiety/depression; Week 24, Level 4: number analyzed (Participants) | 76 | 70
  Anxiety/depression; Week 24, Level 4 | 1 | 2
  Anxiety/depression; Week 24, Level 5: number analyzed (Participants) | 76 | 70
  Anxiety/depression; Week 24, Level 5 | 1 | 0
  Anxiety/depression; Week 32, Level 1: number analyzed (Participants) | 69 | 67
  Anxiety/depression; Week 32, Level 1 | 44 | 54
  Anxiety/depression; Week 32, Level 2: number analyzed (Participants) | 69 | 67
  Anxiety/depression; Week 32, Level 2 | 20 | 11
  Anxiety/depression; Week 32, Level 3: number analyzed (Participants) | 69 | 67
  Anxiety/depression; Week 32, Level 3 | 3 | 2
  Anxiety/depression; Week 32, Level 4: number analyzed (Participants) | 69 | 67
  Anxiety/depression; Week 32, Level 4 | 0 | 0
  Anxiety/depression; Week 32, Level 5: number analyzed (Participants) | 69 | 67
  Anxiety/depression; Week 32, Level 5 | 2 | 0

14. Secondary Outcome: Change From Baseline in EQ-5D-5L Visual Analog Scale (VAS) Score at Weeks 2, 4, 8, 12, 16, 24, and 32
Description: The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome. The EQ-5D-5L questionnaire consists of the following 2 sections: the EQ-5D descriptive system and the EQ Visual Analog Scale (VAS). The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: Level 1 = no problems; Level 2 = slight problems; Level 3 = moderate problems; Level 4 = severe problems; and Level 5 = extreme problems. The EQ VAS records the participant's self-rated health on a vertical VAS (0-100), where the endpoints are labeled "the best health you can imagine" (100 score) and "the worst health you can imagine" (0 score). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 32
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Baseline: number analyzed (Participants) | 89 | 90
  Baseline | 74.21 (18.373) | 73.93 (19.255)
  Change from Baseline at Week 2: number analyzed (Participants) | 81 | 83
  Change from Baseline at Week 2 | 8.85 (18.544) | 4.05 (13.191)
  Change from Baseline at Week 4: number analyzed (Participants) | 81 | 82
  Change from Baseline at Week 4 | 10.73 (19.904) | 5.38 (15.042)
  Change from Baseline at Week 8: number analyzed (Participants) | 80 | 77
  Change from Baseline at Week 8 | 10.75 (19.292) | 6.92 (13.006)
  Change from Baseline at Week 12: number analyzed (Participants) | 76 | 74
  Change from Baseline at Week 12 | 10.82 (20.557) | 8.80 (13.343)
  Change from Baseline at Week 16: number analyzed (Participants) | 75 | 76
  Change from Baseline at Week 16 | 10.97 (20.567) | 7.67 (14.160)
  Change from Baseline at Week 24: number analyzed (Participants) | 72 | 69
  Change from Baseline at Week 24 | 12.22 (21.223) | 10.00 (12.444)
  Change from Baseline at Week 32: number analyzed (Participants) | 67 | 66
  Change from Baseline at Week 32 | 12.34 (21.430) | 11.95 (14.807)

15. Secondary Outcome: Change From Baseline in Quality of Life in Hand Eczema Questionnaire (QOLHEQ) Total Score at Weeks 2, 4, 8, 12, 16, 24, 32, and Follow-up
Description: The QOLHEQ is a validated disease-specific instrument to assess disease-specific health-related quality of life in participants suffering from CHE over the past 7 days. It consists of 30 items that are summarized according to impairments for 4 subscales: symptoms, emotions, limitations in functioning, and treatment and prevention. Each item is scored on a scale of never, rarely, sometimes, often, and all the time. The overall score is calculated by summing all items and ranges from 0 to 117. Higher scores indicate a greater impact on quality of life. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 36
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
scores on a scale
  Baseline: number analyzed (Participants) | 93 | 91
  Baseline | 75.19 (23.864) | 66.52 (23.224)
  Change from Baseline at Week 2: number analyzed (Participants) | 86 | 84
  Change from Baseline at Week 2 | -43.16 (24.337) | -21.98 (18.408)
  Change from Baseline at Week 4: number analyzed (Participants) | 85 | 82
  Change from Baseline at Week 4 | -50.22 (23.579) | -25.10 (21.021)
  Change from Baseline at Week 8: number analyzed (Participants) | 84 | 78
  Change from Baseline at Week 8 | -53.69 (25.377) | -28.44 (22.570)
  Change from Baseline at Week 12: number analyzed (Participants) | 79 | 75
  Change from Baseline at Week 12 | -55.00 (24.109) | -28.95 (24.322)
  Change from Baseline at Week 16: number analyzed (Participants) | 79 | 77
  Change from Baseline at Week 16 | -55.76 (26.741) | -29.56 (25.060)
  Change from Baseline at Week 24: number analyzed (Participants) | 76 | 70
  Change from Baseline at Week 24 | -54.97 (25.757) | -46.60 (24.862)
  Change from Baseline at Week 32: number analyzed (Participants) | 71 | 67
  Change from Baseline at Week 32 | -55.59 (23.885) | -50.04 (24.931)
  Change from Baseline at Safety Follow-up: number analyzed (Participants) | 69 | 67
  Change from Baseline at Safety Follow-up | -48.07 (26.886) | -40.67 (27.454)

16. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire v2.0 in Chronic Hand Dermatitis (WPAI-ChHD) Score at Weeks 2, 4, 8, 12, 16, 24, 32, and Follow-up
Description: The WPAI-ChHD questionnaire is a patient-reported quantitative assessment of the amount of absenteeism (measured as percentage of work time missed [PWTM] due to CHE), presentism, and daily activity impairment (percentage of impairment while working [PIWW] due to CHE, percentage of overall work impairment [POWI] due to CHE, percentage of activity impairment [PAI] due to CHE) attributable to a specific health problem. The WPAI-ChHD is a 6-item questionnaire used to assess the impact of chronic hand dermatitis (ChHD, the same as CHE in this context) on job performance and productivity in the last 7 days. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. Scores range from 0% (no impairment) to 100% (complete impairment). Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to Week 36
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 92
percentage
  PWTM, Baseline: number analyzed (Participants) | 67 | 67
  PWTM, Baseline | 5.68 (16.541) | 2.32 (7.736)
  PWTM, Change from Baseline at Week 2: number analyzed (Participants) | 56 | 58
  PWTM, Change from Baseline at Week 2 | -4.90 (12.817) | -0.90 (5.858)
  PWTM, Change from Baseline at Week 4: number analyzed (Participants) | 57 | 59
  PWTM, Change from Baseline at Week 4 | -3.15 (16.734) | 0.82 (11.469)
  PWTM, Change from Baseline at Week 8: number analyzed (Participants) | 60 | 55
  PWTM, Change from Baseline at Week 8 | -3.92 (19.340) | 0.03 (11.714)
  PWTM, Change from Baseline at Week 12: number analyzed (Participants) | 51 | 54
  PWTM, Change from Baseline at Week 12 | -0.72 (14.356) | -1.40 (9.591)
  PWTM, Change from Baseline at Week 16: number analyzed (Participants) | 51 | 58
  PWTM, Change from Baseline at Week 16 | -0.57 (22.398) | 0.06 (12.294)
  PWTM, Change from Baseline at Week 24: number analyzed (Participants) | 50 | 49
  PWTM, Change from Baseline at Week 24 | -3.09 (12.916) | -0.36 (13.845)
  PWTM, Change from Baseline at Week 32: number analyzed (Participants) | 47 | 41
  PWTM, Change from Baseline at Week 32 | -0.80 (16.359) | -0.83 (15.108)
  PWTM, Change from Baseline at Safety Follow-up: number analyzed (Participants) | 46 | 45
  PWTM, Change from Baseline at Safety Follow-up | -0.23 (9.681) | -0.67 (14.285)
  PIWW, Baseline: number analyzed (Participants) | 69 | 68
  PIWW, Baseline | 46.52 (28.171) | 38.82 (26.176)
  PIWW, Change from Baseline at Week 2: number analyzed (Participants) | 61 | 63
  PIWW, Change from Baseline at Week 2 | -26.56 (26.888) | -12.22 (21.285)
  PIWW, Change from Baseline at Week 4: number analyzed (Participants) | 61 | 62
  PIWW, Change from Baseline at Week 4 | -27.87 (28.642) | -13.87 (21.375)
  PIWW, Change from Baseline at Week 8: number analyzed (Participants) | 63 | 60
  PIWW, Change from Baseline at Week 8 | -32.22 (25.365) | -13.00 (22.944)
  PIWW, Change from Baseline at Week 12: number analyzed (Participants) | 57 | 58
  PIWW, Change from Baseline at Week 12 | -32.81 (27.500) | -11.72 (23.998)
  PIWW, Change from Baseline at Week 16: number analyzed (Participants) | 57 | 60
  PIWW, Change from Baseline at Week 16 | -35.44 (28.162) | -14.33 (20.031)
  PIWW, Change from Baseline at Week 24: number analyzed (Participants) | 54 | 54
  PIWW, Change from Baseline at Week 24 | -32.96 (27.584) | -28.52 (24.984)
  PIWW, Change from Baseline at Week 32: number analyzed (Participants) | 49 | 48
  PIWW, Change from Baseline at Week 32 | -35.51 (26.775) | -30.21 (24.796)
  PIWW, Change from Baseline at Safety Follow-up: number analyzed (Participants) | 50 | 48
  PIWW, Change from Baseline at Safety Follow-up | -30.20 (30.672) | -21.67 (23.730)
  POWI, Baseline: number analyzed (Participants) | 67 | 67
  POWI, Baseline | 47.82 (28.060) | 40.02 (26.651)
  POWI, Change from Baseline at Week 2: number analyzed (Participants) | 56 | 58
  POWI, Change from Baseline at Week 2 | -27.50 (26.315) | -10.85 (20.548)
  POWI, Change from Baseline at Week 4: number analyzed (Participants) | 57 | 59
  POWI, Change from Baseline at Week 4 | -25.78 (28.135) | -11.08 (22.539)
  POWI, Change from Baseline at Week 8: number analyzed (Participants) | 60 | 55
  POWI, Change from Baseline at Week 8 | -32.66 (25.633) | -10.82 (21.500)
  POWI, Change from Baseline at Week 12: number analyzed (Participants) | 51 | 54
  POWI, Change from Baseline at Week 12 | -32.55 (29.872) | -11.99 (25.552)
  POWI, Change from Baseline at Week 16: number analyzed (Participants) | 51 | 58
  POWI, Change from Baseline at Week 16 | -33.67 (30.196) | -14.10 (21.897)
  POWI, Change from Baseline at Week 24: number analyzed (Participants) | 50 | 49
  POWI, Change from Baseline at Week 24 | -33.95 (29.526) | -28.35 (29.678)
  POWI, Change from Baseline at Week 32: number analyzed (Participants) | 47 | 41
  POWI, Change from Baseline at Week 32 | -34.73 (28.130) | -29.59 (29.227)
  POWI, Change from Baseline at Safety Follow-up: number analyzed (Participants) | 46 | 45
  POWI, Change from Baseline at Safety Follow-up | -29.88 (32.391) | -21.20 (26.726)
  PAI, Baseline: number analyzed (Participants) | 89 | 91
  PAI, Baseline | 56.40 (26.079) | 49.45 (24.466)
  PAI, Change from Baseline at Week 2: number analyzed (Participants) | 81 | 84
  PAI, Change from Baseline at Week 2 | -30.37 (26.667) | -11.43 (21.236)
  PAI, Change from Baseline at Week 4: number analyzed (Participants) | 81 | 82
  PAI, Change from Baseline at Week 4 | -34.81 (26.651) | -16.71 (22.611)
  PAI, Change from Baseline at Week 8: number analyzed (Participants) | 80 | 78
  PAI, Change from Baseline at Week 8 | -36.25 (26.259) | -17.18 (24.169)
  PAI, Change from Baseline at Week 12: number analyzed (Participants) | 76 | 75
  PAI, Change from Baseline at Week 12 | -39.21 (26.671) | -20.13 (27.680)
  PAI, Change from Baseline at Week 16: number analyzed (Participants) | 75 | 77
  PAI, Change from Baseline at Week 16 | -41.07 (27.439) | -18.70 (22.381)
  PAI, Change from Baseline at Week 24: number analyzed (Participants) | 72 | 70
  PAI, Change from Baseline at Week 24 | -38.47 (27.304) | -35.71 (26.842)
  PAI, Change from Baseline at Week 32: number analyzed (Participants) | 68 | 67
  PAI, Change from Baseline at Week 32 | -39.12 (25.553) | -38.36 (25.382)
  PAI, Change from Baseline at Safety Follow-up: number analyzed (Participants) | 68 | 67
  PAI, Change from Baseline at Safety Follow-up | -32.06 (27.782) | -26.27 (28.542)

17. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) in the DBVC Period
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up.
Time Frame: up to Week 16
Population: Safety Population: all randomized participants who applied study treatment at least once. Treatment groups were determined according to the actual treatment the participant applied on Day 1 regardless of assigned study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) to chronic hand eczema (CHE) lesions on the hands and wrists (if applicable) for 16 weeks.
- DBVC Period: Vehicle Cream BID: Participants applied matching vehicle cream BID to CHE lesions on the hands and wrists (if applicable) for 16 weeks.
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 94 | 92
Participants | 36 | 29

18. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE in the DBVC Period
Description: A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up. The severity of AEs was based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 using Grades 1 through 5. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to Week 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 94 | 92
Participants | 2 | 1

19. Secondary Outcome: Number of Participants With Any TEAE in the OLE Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up.
Time Frame: up to Week 36
Population: Open-label Evaluable Population: all participants who applied study treatment at least once during the OLE Period
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied ruxolitinib 1.5% cream BID during the DBVC Period continued to apply ruxolitinib 1.5% cream BID as needed for an additional 16 weeks in the OLE Period.
- OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID: Participants who completed the Week 16 assessments with no safety concerns could continue into the 16-week OLE Period. Participants who applied vehicle cream BID during the DBVC Period applied ruxolitinib 1.5% cream BID as needed for 16 weeks in the OLE Period.
Arm/Group | Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 77
Participants | 10 | 25

20. Secondary Outcome: Number of Participants With Any ≥Grade 3 TEAE in the OLE Period
Description: as for outcome 18
Time Frame: up to Week 36
Population: Open-label Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 77
Participants | 1 | 1

21. Secondary Outcome: Number of Participants With Clinically Meaningful Changes or Trends in Laboratory (Hematology and Serum Chemistry) Parameters or Vital Signs in the DBVC Period
Description: The investigator determined whether a change was clinically meaningful.
Time Frame: up to Week 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind, Vehicle-Controlled (DBVC) Period: Ruxolitinib 1.5% Cream BID | DBVC Period: Vehicle Cream BID
Number analyzed (Participants) | 94 | 92
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Meaningful Changes or Trends in Laboratory (Hematology and Serum Chemistry) Parameters or Vital Signs in the OLE Period
Description: The investigator determined whether a change was clinically meaningful.
Time Frame: up to Week 36
Population: Open-label Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Extension (OLE) Period: Ruxolitinib 1.5% Cream BID | OLE Period: Vehicle Cream to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 77
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Week 36
Description: For participants who were on vehicle up to Week 16 and then switched to ruxolitinib, AEs are presented by the treatment they were on at the onset of the event.
Groups:
- Vehicle Cream BID: Participants applied matching vehicle cream twice daily (BID) to chronic hand eczema (CHE) lesions on the hands and wrists (if applicable) for 16 weeks.
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream BID to CHE lesions on the hands and wrists (if applicable) for 16 weeks in the DBVC Period and for 16 weeks in the OLE Period. Participants who applied matching vehicle cream BID to CHE for 16 weeks during the DBVC Period and completed the Week 16 assessments with no safety concerns applied ruxolitinib 1.5% cream for 16 weeks during the OLE Period.
Arm/Group | Vehicle Cream BID | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/92 | 1/171
Serious Adverse Events (participants affected / at risk) | 1/92 | 5/171
Other Adverse Events (participants affected / at risk) | 9/92 | 10/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=92) | Ruxolitinib 1.5% Cream BID (N=171)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=92) | Ruxolitinib 1.5% Cream BID (N=171)
Nasopharyngitis (Infections and infestations) | 9 (10) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT05906628/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT05906628/SAP_001.pdf